CLINICAL TRIAL: NCT05978739
Title: A Randomized,Open-label, Multicenter, Phase II Trial Evaluating Two Different Doses of Orelabrutinib in Mantle Cell Lymphoma
Brief Title: Evaluating Different Doses of Orelabrutinib in MCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: InnoCare Pharma Inc. (Industry)
Collaborators: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00127
Record Dates: First submitted 2023-07-11; First posted 2023-08-07 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — orelabrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orelabrutinib high dose (Experimental)
  Interventions: Drug: Orelabrutinib High dose
- Orelabrutinib low dose (Experimental)
  Interventions: Drug: Orelabrutinib Low dose

INTERVENTIONS:
Drug: Orelabrutinib High dose — Orelabrutinib will be administered as 3 tablets once per day
  Arms: Orelabrutinib high dose
Drug: Orelabrutinib Low dose — Orelabrutinib will be administered as 1 tablet once per day
  Arms: Orelabrutinib low dose

SUMMARY:
This is A Randomized,Open-label, Multicenter, Phase II Trial Evaluating Two Different Doses of Orelabrutinib in Mantle Cell Lymphoma to Evaluate the Efficacy and Safety in Mantle Cell Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥ 18 years of age.
2. Mantle cell lymphoma (MCL) confirmed by histopathology.
3. Subjects who have not previously received standard systemic care and relapsing/refractory subjects who have previously received standard systemic care.
4. At least one measurable lesion.
5. ECOG Physical fitness score 0-2 points.
6. Expected survival time ≥ 4 months.
7. Full hematology function.
8. Blood clotting function is basically normal.
9. Subjects with basically normal liver, kidney and heart function.
10. Subject voluntarily signs a written ICF.
11. The serum pregnancy test of female subjects with fertility potential was negative within 7 days before the first dosing.
12. Female subjects with reproductive potential or male subjects and their partners must agree to use effective contraception for at least 6 months from signing the ICF until the last dose of the study drug.

Exclusion Criteria:

1. Adequate treatment with BTK inhibitors.
2. Have a history of severe allergic disease and a history of severe drug allergy.
3. Subjects who have received the treatment or drug restricted in the protocol within the time specified for the first use of the investigational drug.
4. The last use of a potent CYP3A inhibitor or potent CYP3A inducer (including food, western medicine, and Chinese medicine) was less than 2 weeks (or less than 5 half-lives, depending on the time) from the first trial, or plan to take a potent CYP3A inhibitor or potent CYP3A inducer drug or food during the study period.
5. History of other active malignant diseases within 2 years prior to screening.
6. Subjects with systemic bacterial, viral, fungal (other than nail fungal infections) or parasitic infections with poorly controlled activity.
7. Indicates active hepatitis B or C virus infection.
8. There are diseases that are excluded from the criteria in the programme.
9. Toxicity of previous anticancer therapy was still ≥ grade 2 at the start of study therapy (according to CTCAE V5.0).
10. History of severe bleeding disorder.
11. People with a known history of alcohol or drug abuse.
12. Subjects with mental disorders or poor compliance.
13. Pregnant or lactating female subjects.
14. Other conditions deemed unsuitable for participation in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
Objective response rate（ORR） | Through study completion, an average of 2 year
  Proportion of subjects with tumor response of Complete Response（CR） or Partial Response（PR） after treatment in total subjects.

SECONDARY OUTCOMES:
Complete Response Rate （CRR） | Through study completion, an average of 2 year
  The proportion of subjects with tumor response of Complete Response（CR） after treatment in total subjects.
Progression-Free Survival (PFS) | Through study completion, an average of 2 year
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first.
Duration of Response (DoR) | Through study completion, an average of 2 year
  The time from documentation of objective response to the first occurrence of tumor progression or death due to any cause, whichever occurs first.
Maximum concentration (Cmax,ss) | Predose up to 24 hours postdose
Time to maximum concentration (Tmax) | Predose up to 24 hours postdose
Area under the plasma concentration-time curve (AUC) | Predose up to 24 hours postdose
Half-life (T1/2) | Predose up to 24 hours postdose
Apparent clearance (CL/F) | Predose up to 24 hours postdose
Adverse events（AEs） | Through study completion, an average of 2 year
Serious adverse events （SAEs） | Through study completion, an average of 2 year

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Sun Yat-sen University Cancer Center, Guangdong, Guangzhou
  - Nanyang Second General Hospital, Nanyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Chenzhou First People's Hospital, Chenzhou, Hunan
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - The Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Uygur Autonomous Region
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang